CLINICAL TRIAL: NCT02295098
Title: Comparison of Epidural and Paracostal Catheter Placement for Pain Control After Rib Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-1979
Record Dates: First submitted 2014-11-09; First posted 2014-11-20 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Rib Fractures; Wounds and Injuries
MeSH Terms: conditions — Rib Fractures; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic epidural catheter (Active Comparator): Thoracic epidurals work by delivering local anesthetics and narcotics to the epidural space, which then diffuse into the spinal nerve roots and block the transmission of pain from the chest wall to the spinal cord and brain.
  Interventions: Other: Thoracic epidural catheter placement
- Paracostal catheter (Active Comparator): Paracostal catheters run along the outer surface of the chest wall and act by delivering local anesthetics to the intercostal nerves as traverse the lower border of the ribs.
  Interventions: Other: Paracostal catheter placement

INTERVENTIONS:
Other: Thoracic epidural catheter placement — Thoracic epidurals work by delivering local anesthetics and narcotics to the epidural space, which then diffuse into the spinal nerve roots and block the transmission of pain from the chest wall to the spinal cord and brain.
  Arms: Thoracic epidural catheter
Other: Paracostal catheter placement — Paracostal catheters run along the outer surface of the chest wall and act by delivering local anesthetics to the intercostal nerves as traverse the lower border of the ribs.
  Arms: Paracostal catheter

SUMMARY:
The investigators plan to compare the incidence of successful placement of epidural pain catheters versus paracostal catheters for the control of pain and prevention of pulmonary complications for adult trauma patients with blunt chest wall trauma resulting in multiple rib fractures. When a trauma patient has > or = to 3 rib fractures on the same side, is being admitted to the Surgical ICU, and is encountered within 72 hours from the time of their injury, they will be eligible for the study. If they (or a proxy) choose to participate, consent will be obtained and they will randomly be assigned to receive either an epidural or paracostal catheter for pain control. The aim of the study is to determine if paracostal catheters are noninferior to epidurals for controlling pain in multisystem trauma patients. Secondarily the investigators will evaluate success and time of placement of the assigned intervention and follow the patient throughout their hospital course to compare the success of analgesia provided by each modality along with any complications and/or benefits of the two types of catheters.

ELIGIBILITY:
Inclusion Criteria:

* >/= 3 rib fractures on a single side
* Admitted to the Surgical ICU
* Recruited within 24 hours of admission

Exclusion Criteria:

* Patient allergy to local anesthetics
* Patient refusal
* Inability to consent for any reason
* Prisoners
* Age < 18
* Pregnant women (pregnancy screen performed as part of routine trauma admission labs)
* Absolute contraindications for either thoracic epidural or paracostal pain catheter placement which include:

  1. Localized rash or skin infection over the likely site of insertion (We never want to translocate infectious material from the skin to the epidural space or even into the soft tissue where paracostal catheters lay, although for these there is more flexibility in adjusting placement)
  2. Spinal/vertebral instability/fracture including any significant vertebral body injury and 3 or more spinous process fractures near the level of desired epidural placement (transverse process fractures are not considered a contraindication)
  3. History of extensive back surgery at the level of desired epidural placement
  4. Severe aortic stenosis, mitral stenosis, or pulmonary hypertension
  5. Inability to correct coagulopathy (to International Normalized Ratio>1.5)
  6. Persistent hemodynamic instability (hypotension with Systolic Blood Pressure<90 that does not respond to initial fluid boluses and requires ongoing pressors beyond the 72 hour window for enrollment)
  7. Inability to cooperate and participate in placement (if intubated and sedated, for example) or to lie in the correct position for placement (lateral decubitus for paracostal pain catheters, either sitting up or lateral decubitus for epidural placement)
  8. Concern for elevated intracranial pressure (we imagine these patients will also be intubated)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08-19 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Pain assessment immediately before and after catheter placement | within an hour before and after catheter placement
  Pain scores are assessed by nursing on an hourly basis in the ICU

SECONDARY OUTCOMES:
successful placement of randomized intervention (paracostal vs. epidural catheter) | Within 24 hours of recruitment
Comparison of analgesic effect as measured by daily pain scores | Duration of admission up to 30 days
  Daily pain scores are assessed by nursing hourly in the ICU and every shift after transfer to the floor. These are measured by the Critical-Care Pain Observation Tool (CPOT).
Comparison of improvements in pulmonary function | Duration of admission up to 30 days as long as the patient remains in the ICU
  Respiratory therapist assessment of pulmonary function (including incentive spirometry maximum, forced vital capacity, peak expiratory flow, respiratory rate and supplemental oxygen requirement) every shift will be reviewed for evidence of respiratory embarrassment.
Comparison of improvements in maximum daily incentive spirometry | Duration of admission up to 30 days
  Nursing assessment of incentive spirometry every shift will be reviewed for evidence of respiratory embarrassment.
Comparison of improvements in forced vital capacity | Duration of admission up to 30 days as long as the patient remains in the ICU
  Respiratory therapist assessment of forced vital capacity every shift will be reviewed for evidence of respiratory embarrassment.
Comparison of improvements in peak expiratory flow | Duration of admission up to 30 days as long as the patient remains in the ICU
  Respiratory therapist assessment of peak expiratory flow every shift will be reviewed for evidence of respiratory embarrassment.
Number of patients in each group with pulmonary complications | Duration of admission up to 30 days
  All patients will be assessed daily for other evidence of respiratory embarrassment including: hypoxemia, pneumonia, empyema, need for mechanical ventilation, or readmission due to pulmonary complaints.
ICU length of stay | Duration of admission up to 30 days
Hospital length of stay | Duration of admission up to 30 days
30-day Mortality | Duration of admission up to 30 days
Comparison of daily requirement for narcotics and other additional pain medications. | Duration of admission up to 30 days
Number of patients who had alterations in their care related to the studied interventions (paracostal vs. epidural catheters) | Duration of admission up to 30 days
  We will assess any possible alterations in care related to interventions (e.g., failure to mobilize, anticoagulate, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Nina E Glass, MD, Principal Investigator — Denver Health Medical Center, Department of Surgery, University of Colorado, Denver
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Simon BJ, Cushman J, Barraco R, Lane V, Luchette FA, Miglietta M, Roccaforte DJ, Spector R; EAST Practice Management Guidelines Work Group. Pain management guidelines for blunt thoracic trauma. J Trauma. 2005 Nov;59(5):1256-67. doi: 10.1097/01.ta.0000178063.77946.f5. No abstract available. PMID 16385313
- [Background] Truitt MS, Mooty RC, Amos J, Lorenzo M, Mangram A, Dunn E. Out with the old, in with the new: a novel approach to treating pain associated with rib fractures. World J Surg. 2010 Oct;34(10):2359-62. doi: 10.1007/s00268-010-0651-9. PMID 20567973
- [Background] Sirmali M, Turut H, Topcu S, Gulhan E, Yazici U, Kaya S, Tastepe I. A comprehensive analysis of traumatic rib fractures: morbidity, mortality and management. Eur J Cardiothorac Surg. 2003 Jul;24(1):133-8. doi: 10.1016/s1010-7940(03)00256-2. PMID 12853057
- [Background] Moon MR, Luchette FA, Gibson SW, Crews J, Sudarshan G, Hurst JM, Davis K Jr, Johannigman JA, Frame SB, Fischer JE. Prospective, randomized comparison of epidural versus parenteral opioid analgesia in thoracic trauma. Ann Surg. 1999 May;229(5):684-91; discussion 691-2. doi: 10.1097/00000658-199905000-00011. PMID 10235527
- [Background] Holcomb JB, McMullin NR, Kozar RA, Lygas MH, Moore FA. Morbidity from rib fractures increases after age 45. J Am Coll Surg. 2003 Apr;196(4):549-55. doi: 10.1016/S1072-7515(02)01894-X. PMID 12691929
- [Background] Ho AM, Karmakar MK, Critchley LA. Acute pain management of patients with multiple fractured ribs: a focus on regional techniques. Curr Opin Crit Care. 2011 Aug;17(4):323-7. doi: 10.1097/MCC.0b013e328348bf6f. PMID 21716105
- [Background] Grider JS, Mullet TW, Saha SP, Harned ME, Sloan PA. A randomized, double-blind trial comparing continuous thoracic epidural bupivacaine with and without opioid in contrast to a continuous paravertebral infusion of bupivacaine for post-thoracotomy pain. J Cardiothorac Vasc Anesth. 2012 Feb;26(1):83-9. doi: 10.1053/j.jvca.2011.09.003. Epub 2011 Nov 17. PMID 22100213
- [Background] Gebhardt R, Mehran RJ, Soliz J, Cata JP, Smallwood AK, Feeley TW. Epidural versus ON-Q local anesthetic-infiltrating catheter for post-thoracotomy pain control. J Cardiothorac Vasc Anesth. 2013 Jun;27(3):423-6. doi: 10.1053/j.jvca.2013.02.017. PMID 23672860
- [Background] Dahlgren N, Tornebrandt K. Neurological complications after anaesthesia. A follow-up of 18,000 spinal and epidural anaesthetics performed over three years. Acta Anaesthesiol Scand. 1995 Oct;39(7):872-80. doi: 10.1111/j.1399-6576.1995.tb04190.x. PMID 8848884
- [Background] Carrier FM, Turgeon AF, Nicole PC, Trepanier CA, Fergusson DA, Thauvette D, Lessard MR. Effect of epidural analgesia in patients with traumatic rib fractures: a systematic review and meta-analysis of randomized controlled trials. Can J Anaesth. 2009 Mar;56(3):230-42. doi: 10.1007/s12630-009-9052-7. Epub 2009 Feb 11. PMID 19247744
- [Background] Bulger EM, Edwards T, Klotz P, Jurkovich GJ. Epidural analgesia improves outcome after multiple rib fractures. Surgery. 2004 Aug;136(2):426-30. doi: 10.1016/j.surg.2004.05.019. PMID 15300210
- [Background] Bulger EM, Arneson MA, Mock CN, Jurkovich GJ. Rib fractures in the elderly. J Trauma. 2000 Jun;48(6):1040-6; discussion 1046-7. doi: 10.1097/00005373-200006000-00007. PMID 10866248
- [Background] Brasel KJ, Guse CE, Layde P, Weigelt JA. Rib fractures: relationship with pneumonia and mortality. Crit Care Med. 2006 Jun;34(6):1642-6. doi: 10.1097/01.CCM.0000217926.40975.4B. PMID 16625122
- [Result] Mohta M, Verma P, Saxena AK, Sethi AK, Tyagi A, Girotra G. Prospective, randomized comparison of continuous thoracic epidural and thoracic paravertebral infusion in patients with unilateral multiple fractured ribs--a pilot study. J Trauma. 2009 Apr;66(4):1096-101. doi: 10.1097/TA.0b013e318166d76d. PMID 19359920
- [Result] Truitt MS, Murry J, Amos J, Lorenzo M, Mangram A, Dunn E, Moore EE. Continuous intercostal nerve blockade for rib fractures: ready for primetime? J Trauma. 2011 Dec;71(6):1548-52; discussion 1552. doi: 10.1097/TA.0b013e31823c96e0. PMID 22182865